CLINICAL TRIAL: NCT00290147
Title: An Open-Label, Dose Escalation, Phase I Safety, and Immunogenicity Trial of a Dengue Serotype 1 (DEN-1) Premembrane (prM) and Envelope (E) DNA Vaccine (D1ME100) in Healthy Adults Volunteers
Brief Title: Safety and Immunogenicity Study of a Dengue Virus DNA Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: United States Army Medical Materiel Development Activity (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NMRC 2004.0002; WRAIR 1191 (Other: WRAIR ID); HSRRB A-13304 (Other: IRB); 62787A 810S A0235 (Other)
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Dengue
Keywords: Dengue; DNA vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1.0 mg of D1ME100 vaccine (Experimental): 1.0 mg dose of DME100 vaccine delivered by Biojector IM injections at 0, 1 and 5 months
  Interventions: Biological: D1ME100 (dengue-1 premembrane/envelope DNA vaccine)
- 5.0 mg of D1ME100 vaccine (Experimental): 5.0 mg dose of DME100 vaccine delivered by Biojector IM injections at 0, 1 and 5 months
  Interventions: Biological: D1ME100 (dengue-1 premembrane/envelope DNA vaccine)

INTERVENTIONS:
Biological: D1ME100 (dengue-1 premembrane/envelope DNA vaccine) — IM injection delivered by Biojector

SUMMARY:
The purpose of this study is to exame the safety of a DNA vaccine against dengue-1.

DETAILED DESCRIPTION:
Dengue is a desease that affects 100 million people throughout the world mainly in tropical countries in the South Pacific, Asia, the Caribbean, and Africa. The disease often presents with high fever, severe headache, and joint/muscle pain that usually goes away on its own, but it can also present as a sometimes deadly hemorrhagic (bleeding) disease. Humans catch this disease by being bitten by mosquitoes that have been infected with dengue virus. Scientists at the Naval Medical Research Center have been working on vaccines to prevent dengue disease. This vaccine, referred to as D1ME, is an experimental DNA vaccine that contains genes from the dengue-1 virus. The purpose of this study is to test the safety of a new experimental vaccine against dengue and to see if the vaccine can stimulate the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Available to participate for the duration of the study (approximately 12 months)
* Completion and review of knowledge assement quiz

Exclusion Criteria:

* Pregnant (by history or as ascertained by pregnancy test) or lactating female
* Female who intends to become pregnant during the study
* Plan to have elective surgery during the study period
* HIV infection
* Known immunodeficiency or currently receiving immunosuppressive therapy (inhaled and topical steroids are allowed)
* History of splenectomy
* Administration of a vaccine not foreseen by the study protocol during the period starting 30 days before each dose of vaccine and ending 30 days after vaccination
* Evidence of active (acute or chronic) hepatitis B or C infection
* Autoimmune diseaseor subjects who describe a first-degree relative with clearly documented autoimmune disease
* Acute or chronic, clinically significant cardiac, pulmonary, hepatic, or renal abnormality, as determined by physical examination or basic laboratory screening
* Clinical or laboratory evidence of significant anemia
* History of flavivirus infection or previous receipt of flavivirus vaccine
* Positive serology for flaviviruses (all four dengue virus serotypes, Japanese encephalitis, Yellow fever virus, and West Nile virus), HIV-1, Hepatitis B surface antigen, or anti-hepatitis C virus antibodies prior to enrollment
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 60 days preceding the first dose of study vaccine, or planned use during the study period.
* Previous history of allergic or anaphylactic reaction to any vaccine
* Planned travel to areas with endemic dengue during the study period
* Any other significant finding which, in the opinion of the investigator, would increase the risk of having an adverse outcome from participating in this protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2006-01; Primary Completion 2006-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charmagne Beckett, MD, Principal Investigator — Naval Medical Research Center
Locations (1):
- Walter Reed Army Institute of Research, Bldg 503, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danko JR, Kochel T, Teneza-Mora N, Luke TC, Raviprakash K, Sun P, Simmons M, Moon JE, De La Barrera R, Martinez LJ, Thomas SJ, Kenney RT, Smith L, Porter KR. Safety and Immunogenicity of a Tetravalent Dengue DNA Vaccine Administered with a Cationic Lipid-Based Adjuvant in a Phase 1 Clinical Trial. Am J Trop Med Hyg. 2018 Mar;98(3):849-856. doi: 10.4269/ajtmh.17-0416. Epub 2018 Jan 18. PMID 29363446
- [Derived] Beckett CG, Tjaden J, Burgess T, Danko JR, Tamminga C, Simmons M, Wu SJ, Sun P, Kochel T, Raviprakash K, Hayes CG, Porter KR. Evaluation of a prototype dengue-1 DNA vaccine in a Phase 1 clinical trial. Vaccine. 2011 Jan 29;29(5):960-8. doi: 10.1016/j.vaccine.2010.11.050. Epub 2010 Nov 25. PMID 21111785

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 healthy adult volunteers enrolled to participate at the Naval Medical Research Center site
Period: Overall Study
Arm/Group | 1.0 mg of D1ME100 Vaccine | 5.0 mg of D1ME100 Vaccine
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.0 mg of D1ME100 Vaccine | 5.0 mg of D1ME100 Vaccine | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (8.60) | 36.9 (9.89) | 38.5 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 6 | 9 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 1 | 2 | 3
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 22
Active Duty Military [Count of Participants; unit: Participants] | 0 | 2 | 2
Civilian [Count of Participants; unit: Participants] | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Systemic and Local Reactogenicity Rates for Ungraded Symptoms
Description: Summary of ungraded systemic and local reactogenicity symptoms following each vaccination
Time Frame: Months 0, 1 and 5
Measure: Count of Participants; unit: Participants
Arm/Group | 1.0 mg of D1ME100 Vaccine | 5.0 mg of D1ME100 Vaccine
Number analyzed (Participants) | 10 | 12
Participants
  Systemic: Fever | 0 | 1
  Systemic: Chills | 0 | 2
  Systemic: Rash | 0 | 0
  Systemic: Loss of Appetite | 0 | 2
  Systemic: Red Eyes | 1 | 0
  Local: Redness at Vaccine Site | 0 | 5

2. Secondary Outcome: Anti-dengue Antibody and T-cell and B-cell Responders
Description: Number of participants who responded, are reported. Response or a positive ELISPOT assay was defined as >65 spot forming cells per million PBMC for T-cells and >20 spot forming cells per million PBMC for B-cells
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1.0 mg of D1ME100 Vaccine | 5.0 mg of D1ME100 Vaccine
Number analyzed (Participants) | 9 | 12
Participants
  B-Cell : All | 4 | 7
  B-Cell : DEN-1 | 4 | 6
  B-Cell : DEN-2 | 4 | 2
  B-Cell : DEN-3 | 4 | 7
  B-Cell : DEN-4 | 3 | 8
  T-Cell : All | 5 | 11
  T-Cell : DEN-1 | 5 | 11
  T-Cell : DEN-2 | 2 | 6
  T-Cell : DEN-3 | 2 | 6
  T-Cell : DEN-4 | 1 | 7

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | 1.0 mg of D1ME100 Vaccine | 5.0 mg of D1ME100 Vaccine
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/12
Other Adverse Events (participants affected / at risk) | 10/10 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.0 mg of D1ME100 Vaccine (N=10) | 5.0 mg of D1ME100 Vaccine (N=12)
Alcohol withdrawal (Psychiatric disorders) | 0 (0) | 1 (1) — Not related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1.0 mg of D1ME100 Vaccine (N=10) | 5.0 mg of D1ME100 Vaccine (N=12)
Malaise (General disorders) | 1 (1) | 0 (0) — Severe; Not related
Tenderness (General disorders) | 10 (12) | 12 (20) — Mild; Probable
Echymosis right arm following trauma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Mild; Not related
Right arm pain following trauma (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Mild; Not related
Malaise (General disorders) | 2 (2) | 1 (1) — Moderate; Unlikely related
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) — Moderate; Not related
Malaise (General disorders) | 2 (2) | 1 (1) — Mild; Unlikely related
Seasonal allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Mild; Not related
Chest pain following trauma (General disorders) | 1 (1) | 0 (0) — Mild; Not related
Jaw pain following trauma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Mild; Not related
Elevated CPK (Investigations) | 3 (3) | 1 (1) — Severe; Unlikely related
Low blood sugar (Investigations) | 1 (1) | 0 (0) — Mild; Not related
Elevated CPK (Investigations) | 7 (7) | 2 (2) — Mild; Unlikely related
Elevated CPK (Investigations) | 2 (2) | 5 (5) — Moderate; Unlikely related
Decreased bicarbonate level (Investigations) | 2 (2) | 0 (0) — Mild; Unlikely related
Increased diastolic BP (Investigations) | 1 (1) | 2 (2) — Mild; Not related
Burn left hand following trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Mild; Not related
Increased systolic BP (Investigations) | 1 (1) | 3 (3) — Mild; Not related
Urine - Trace protein (Investigations) | 1 (1) | 0 (0) — Mild; Not related
Elevated eosinophilis (Investigations) | 1 (1) | 0 (0) — Mild; Unlikely related
Decreased HgB (Investigations) | 1 (1) | 0 (0) — Mild; Not related
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) — Mild; Unlikely related
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) — Mild; Unlikely related
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Mild; Not related
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Mild; Unlikely related
Right shoulder discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Mild; Unlikely related
Elevated CK (Investigations) | 1 (1) | 0 (0) — Severe; Unlikely related
Elevated CPK (Investigations) | 1 (1) | 0 (0) — Mild; Not related
Tenderness (General disorders) | 2 (2) | 1 (1) — Moderate; Probable
Nausea (Gastrointestinal disorders) | 1 (1) | 2 — Mild; Not related
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) — Mild; Not related
Flu illness (General disorders) | 1 (1) | 0 (0) — Moderate; Not related
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Mild; Not related
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) — Moderate; Not related
Right lower wisdom tooth pain / impaction (Gastrointestinal disorders) | 1 (1) | 0 (0) — Moderate; Not related
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) — Mild; Not related
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) — Mild; Not related
Intermittent left arm pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Moderate; Unlikely related
Intermittent left arm weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Moderate; Unlikely related
Black out (syncope) episode (Nervous system disorders) | 1 (1) | 0 (0) — Moderate; Not related
Herpes zoster (shingles) (Infections and infestations) | 1 (1) | 0 (0) — Moderate; Not related
Elevated calcium (Investigations) | 1 (1) | 0 (0) — Mild; Not related
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) — Mild; Probable
Malaise (General disorders) | 1 (1) | 0 (0) — Mild; Probable
Induration (General disorders) | 1 (1) | 8 (8) — Mild; Probable
Elevated systolic BP (Investigations) | 0 (0) | 4 (4) — Mild; Unlikely related
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Severe; Unlikely related
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Moderate; Suspected
Photophobia (Eye disorders) | 0 (0) | 1 (1) — Moderate; Suspected
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Mild; Unlikely related
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Moderate; Suspected
Headache (Nervous system disorders) | 0 (0) | 2 (2) — Moderate; Unlikely related
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) — Mild; Unlikely related
Headache (Nervous system disorders) | 0 (0) | 7 (7) — Mild; Unlikely related
Photophobia (Eye disorders) | 0 (0) | 2 (2) — Mild; Unlikely related
Flu-like syndrome (fever, chills) (General disorders) | 0 (0) | 1 (1) — Moderate; Unlikely related
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 12 (12) — Mild; Probable
Increased respiratory rate (Investigations) | 0 (0) | 3 (3) — Mild; Not related
Loss of taste (Nervous system disorders) | 0 (0) | 1 (1) — Mild; Probable
Malaise (General disorders) | 0 (0) | 3 (3) — Mild; Suspected
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Mild; Suspected
Papule (skin lesion) at vaccination site (General disorders) | 0 (0) | 1 (1) — Mild; Suspected
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Mild; Suspected
Cold (Infections and infestations) | 0 (0) | 1 (1) — Mild; Not related
Burn on left ankle (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Mild; Not related
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Moderate; Not related
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Moderate; Not related
Headache (Nervous system disorders) | 0 (0) | 3 (3) — Mild; Not related
Trace proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) — Mild; Unlikely related
Toothache (Gastrointestinal disorders) | 0 (0) | 4 (4) — Mild; Not related
Tooth infection (Infections and infestations) | 0 (0) | 2 (2) — Mild; Not related
Eye pain (Eye disorders) | 0 (0) | 1 (1) — Mild; Suspected
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Mild; Not related
Weird dreams (nightmares) (Psychiatric disorders) | 0 (0) | 1 (1) — Mild; Not related
Malaise (General disorders) | 0 (0) | 1 (1) — Moderate; Suspected
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Mild; Unlikely related
Left forearm injury and pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Mild; Not related
Decreased WBC - 3.3 (Investigations) | 0 (0) | 2 (2) — Mild; Not related
Elevated systolic BP (142) (Investigations) | 0 (0) | 1 (1) — Mild; Not related
Decreased lymphocytes (818) (Investigations) | 0 (0) | 1 (1) — Mild; Not related
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) — Mild; Not related
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Mild; Not related
Low WBC (Investigations) | 0 (0) | 1 (1) — Mild; Not related
Low lymphocyte count (Investigations) | 0 (0) | 1 (1) — Mild; Not related
Right knee pain (increased) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Moderate; Not related
Elevated creatinine (Investigations) | 0 (0) | 2 (2) — Moderate; Unlikely related
Elevated creatinine (Investigations) | 0 (0) | 2 (2) — Mild; Unlikely related
Low hemoglobin (Investigations) | 0 (0) | 1 (1) — Mild; Suspected
Mild anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Mild; Unlikely related
Decreased absolute lymphocytes (Investigations) | 0 (0) | 1 (1) — Mild; Not related
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Mild; Not related
Elevated creatine kinase (Investigations) | 0 (0) | 1 (1) — Mild; Unlikely related
Indegestion (Gastrointestinal disorders) | 0 (0) | 1 (1) — Moderate; Not related
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) — Mild; Unlikely related
Elevated DBP (93) (Investigations) | 0 (0) | 1 (1) — Mild; Not related
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) — Mild; Suspected
Elevated diastolic blood pressure (Investigations) | 0 (0) | 2 (2) — Moderate; Not related
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Mild; Suspected
Elevated AST (Investigations) | 0 (0) | 3 (3) — Mild; Not related
Low bicarbonate (Investigations) | 0 (0) | 2 (2) — Mild; Unlikely related
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Mild; Unlikely related
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Moderate; Suspected
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Moderate; Suspected
Elevated diastolic BP (Investigations) | 0 (0) | 1 (1) — Severe; Unlikely related
Elevated systolic BP (Investigations) | 0 (0) | 1 (1) — Moderate; Unlikely related
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Mild; Not related
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Moderate; Suspected
Headache (Nervous system disorders) | 0 (0) | 3 (3) — Mild; Suspected
Decreased CO2 (Investigations) | 0 (0) | 1 (1) — Mild; Not related
Right thigh pain (s/p fall) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Mild; Not related
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Mild; Not related
Chills (General disorders) | 0 (0) | 1 (1) — Mild; Suspected
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Mild; Unlikely related
Trace protein on uA (Investigations) | 0 (0) | 1 (1) — Mild; Unlikely related
Elevated BUN (Investigations) | 0 (0) | 1 (1) — Mild; Not related
Increased CPK (Investigations) | 0 (0) | 1 (1) — Moderate; Unlikely related
Increased HR (109) (Investigations) | 0 (0) | 1 (1) — Mild; Not related
Increased diastolic BP (Investigations) | 0 (0) | 1 (1) — Moderate; Not related
Tooth pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Mild; Not related
Trace proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) — Mild; Not related
Decreased hemoglobin (Investigations) | 0 (0) | 1 (1) — Mild; Not related
Increased respiratory rate - 22 (Investigations) | 0 (0) | 1 (1) — Moderate; Not related
Back ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Mild; Not related
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Mild; Unlikely related
Decreased hemoglobin (Investigations) | 0 (0) | 1 (1) — Mild; Unlikely related
Decreased blood glucose (Investigations) | 0 (0) | 1 (1) — Mild; Not related
Elevated creatinine (Investigations) | 0 (0) | 1 (1) — Mild; Not related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No